CLINICAL TRIAL: NCT02974725
Title: A Phase Ib, Open-label, Multicenter Study of Oral LXH254-centric Combinations in Adult Patients With Advanced or Metastatic KRAS or BRAF Mutant Non-Small Cell Lung Cancer or NRAS Mutant Melanoma
Brief Title: A Phase Ib Study of LXH254-centric Combinations in NSCLC or Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLXH254X2102; 2016-004293-18 (EudraCT Number)
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer; Melanoma
Keywords: NSCLC; Melanoma; NRAS; KRAS; BRAF; LXH254; LTT462; Trametinib; Ribocliclib; Non-small cell lung carcinoma (NSCLC); treatment of lung cancer after first metastasis; lung cancer; lung adenocarcinoma; Large-cell lung carcinoma; Non small cell lung carcinoma; Non small cell lung cancer; Large cell lung carcinoma; Large cell lung cancer; squamous cell lung carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Lung Neoplasms; Adenocarcinoma of Lung | interventions — naporafenib; trametinib; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LXH254+LTT462 (Experimental)
  Interventions: Drug: LXH254; Drug: LTT462
- LXH254+Trametinib (Experimental)
  Interventions: Drug: LXH254; Drug: Trametinib
- LXH254+Ribociclib (Experimental)
  Interventions: Drug: LXH254; Drug: Ribociclib

INTERVENTIONS:
Drug: LXH254 — LXH254 will be supplied as tablet for oral use.
Drug: LTT462 — LTT462 will be supplied as hard gelatin capsule for oral use.
  Arms: LXH254+LTT462
Drug: Trametinib — Trametinib will be supplied as film-coated tablet for oral use
  Arms: LXH254+Trametinib
Drug: Ribociclib — Ribociclib will be supplied in tablets and hard gelatin capsules.
  Arms: LXH254+Ribociclib

SUMMARY:
To characterize safety and tolerability and identify a recommended dose and regimen for the LXH254 in combination with LTT462 or trametinib or ribociclib.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced or metastatic NSCLC or cutaneous melanoma
* Presence of KRAS or BRAF mutation (NSCLC) or NRAS mutation (cutaneous melanoma) in tumor tissue
* All patients participating in this clinical trial must have progressed following standard therapy or, in the opinion of the Investigator, no effective standard therapy exists, is tolerated, appropriate or is considered equivalent to study treatment.
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2

Exclusion Criteria:

-Dose expansion - KRAS or NRAS mutant patients groups: Prior treatment with a RAFi (including any BRAFi and pan-RAFi), MEKi and/or ERKi. (Patients with KRAS mutant NSCLC with prior G12C inhibitor treatments are also excluded in the LXH254+trametinib expansion part). BRAF mutant patients group: Prior treatment with any EGFR, ALK, ROS1, KRAS, RAF (both BRAFV600 selective and pan-RAF), MEK1/2 and/or ERK1/2 inhibitors (for patients with BRAF V600 mutant NSCLC, prior treatments with BRAF and MEK1/2 inhibitors are allowed).

Patients who have received more than 3 lines of anti-cancer therapy are excluded.

* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO.
* Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Patients receiving proton pump inhibitors (PPI) which cannot be discontinued 3 days prior to the start study treatment and for the duration of the study.
* Patients with Gilbert's syndrome or other heritable diseases of bile processing.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) as a measure of safety and tolerability | up to 5 years
Dose limiting toxicities (DLTs) (dose escalation only) | up to 3 years
Tolerability measured by the number of subjects who have interruptions/reductions of study treatment and reason for interruptions/reductions | up to 5 years
Tolerability measured by the dose intensity of study drug, Relative Dose intensity for subjects with non-zero duration of exposure is computed as the ratio of dose intensity and planned dose intentity | Up to 5 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 5 years
Duration of response (DOR) | Up to 5 years
Disease Control Rate (DCR) | Up to 5 years
Progression Free Survival (PFS) | Up to 5 years
Overall Survival (OS) - (dose expansion part only) | Up to 5 years
Derived PK parameter (Cmax) for LXH254 & LTT462: | Up to 5 years
Derived PK parameter (AUC) for LXH254 & LTT462 | Up to 5 years
Changes from baseline of pharmacodynamics (PD) marker DUSP6 in tumor samples | up to 5 years
Derived PK parameter (Cmax) for LXH254 & trametinib | up to 5 years
Derived PK parameter (AUC) for LXH254 & trametinib | Up to 5 years
Derived PK parameter (Cmax) for LXH254 & ribociclib | Up to 5 years
Derived PK parameter (AUC) for LXH254 & ribociclib | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (29):
- United States (6):
  - University of California San Diego ., San Diego, California
  - UCSF Medical Center, San Francisco, California
  - Massachusetts General Hospital SC, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Ctr ., New York, New York
  - Sarah Cannon Research Institute Tennessee Oncology, Nashville, Tennessee
  - Uni of TX MD Anderson Cancer Cntr, Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
- Novartis Investigative Site, Leuven, Belgium
- France (3):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Germany (4):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
- Novartis Investigative Site, Tel Aviv, Israel
- Italy (4):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, Seoul, South Korea
- Spain (5):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Planchard D, Wolf J, Solomon B, Sebastian M, Wermke M, Heist RS, Sun JM, Min Kim T, Reguart N, Sanmamed MF, Felip E, Garrido P, Santoro A, Bootle D, Couillebault XM, Gaur A, Mueller C, Poggio T, Yang J, Moschetta M, Dooms C. A phase Ib study of the combination of naporafenib with rineterkib or trametinib in patients with advanced and metastatic KRAS- or BRAF-mutant non-small cell lung cancer. Lung Cancer. 2024 Nov;197:107964. doi: 10.1016/j.lungcan.2024.107964. Epub 2024 Sep 26. PMID 39383771
- [Derived] de Braud F, Dooms C, Heist RS, Lebbe C, Wermke M, Gazzah A, Schadendorf D, Rutkowski P, Wolf J, Ascierto PA, Gil-Bazo I, Kato S, Wolodarski M, McKean M, Munoz Couselo E, Sebastian M, Santoro A, Cooke V, Manganelli L, Wan K, Gaur A, Kim J, Caponigro G, Couillebault XM, Evans H, Campbell CD, Basu S, Moschetta M, Daud A. Initial Evidence for the Efficacy of Naporafenib in Combination With Trametinib in NRAS-Mutant Melanoma: Results From the Expansion Arm of a Phase Ib, Open-Label Study. J Clin Oncol. 2023 May 10;41(14):2651-2660. doi: 10.1200/JCO.22.02018. Epub 2023 Mar 22. PMID 36947734
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18291